CLINICAL TRIAL: NCT03739229
Title: Reactogenicity, Safety and Immunogenicity of a Live Monovalent А/17/Hong Kong/2017/75108 (H7N9) Influenza Vaccine
Brief Title: Reactogenicity, Safety and Immunogenicity of a LAIV А/17/Hong Kong/2017/75108 H7N9 Influenza Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Research Institute of Influenza, Russia (Other)
Collaborators: World Health Organization (Other); Institute of Experimental Medicine, Russia (Other); Joint Stock Company Microgen, Russia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAIV-H7N9-02
Record Dates: First submitted 2018-11-01; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Vaccine Adverse Reaction
Keywords: pandemic; influenza; vaccine; H7N9
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H7N9 LAIV (Active Comparator): H7N9 live influenza vaccine at study entry (dose 1) and four weeks post-dose one (dose 2), subjects will receive two, 0.25 ml intranasal doses of study vaccine (total dose 0.50 ml at each study vaccine administration).
  Interventions: Biological: Placebo; Biological: H7N9 LAIV
- Placebo (Placebo Comparator): Lyophilized purified allantoic fluid of chicken embryos with stabilizers at study entry (dose 1) and four weeks post-dose one (dose 2), subjects will receive two, 0.25 ml intranasal doses of placebo (total dose 0.50 ml at each placebo administration).
  Interventions: Biological: Placebo; Biological: H7N9 LAIV

INTERVENTIONS:
Biological: Placebo — 2 intranasal administrations of lyophilized purified allantoic fluid of chicken embryos with stabilizers
Biological: H7N9 LAIV — 2 intranasal administrations of H7N9 live influenza vaccine

SUMMARY:
This is a single center phase I, double-blind placebo-controlled study to assess reactogenicity, safety and immunogenicity of a live monovalent A/17/Hong Kong/2017/75108 (H7N9) influenza vaccine in healthy male and female adults, 18 through 49 years of age.

DETAILED DESCRIPTION:
This is a phase I, double-blind, individually-randomized (3:1, vaccine:placebo), controlled trial with two groups, LAIV H7N9 and matched placebo. Healthy male and female adults 18 through 49 years of age will be invited to participate. For feasibility reasons and in order for an independent Safety Monitoring Committee (SMC) to review safety data in a portion of subjects initially, the total cohort of 40 subjects will be enrolled in two cohorts: one cohort of 20 subjects, randomized at 3:1 (15 vaccine and 5 placebo), followed two weeks later by a second identically composed cohort of 20 subjects randomized at 3:1 (15 vaccine and 5 placebo). After all volunteers of the first cohort have been observed for the first isolation period (Day 0 to Day 6) after receipt of dose one, an interim safety review will be performed by a SMC. The SMC will review all AEs and shedding data, for all subjects and will advise if the volunteers of the first cohort may receive dose two of study vaccine or placebo and if the additional 20 volunteers of the second cohort may be enrolled into the study. For each cohort, the procedures and timelines are here summarized.

On the day of first screening (S1), about 7 days (between 4 and 14 days) prior to administration of dose one of study vaccine or placebo, subjects will be screened for eligibility through medical history review, physical examination, testing for serologic evidence of chronic viral infection [human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)], routine biochemical and hematological blood tests and routine urinalysis.

For screening for serologic evidence of chronic viral infections, appropriate pre- and post-test counseling must be provided.

Subject screening for eligibility will continue and be completed on the second screening day (S2). This second screening day will occur the same day as scheduled admission to the isolation unit and administration of study vaccine or placebo (Day 0). Women will undergo pregnancy tests using urine samples. All subjects will undergo an ear, nose and throat (ENT) examination and examination by neurologist. Fully eligible subjects will be admitted to the isolation unit. At that time, nasal swabs, nasal wick, saliva and blood specimens will be collected for virologic and immunological testing prior to administration of study vaccine or placebo. Blood and urine specimens will be again collected for routine biochemical and hematological blood tests and urinanalysis; these results will serve to define baseline status for subject prior to receipt of study vaccine or placebo but will not be used for screening purposes. Subjects and investigators conducting assessments of safety will be unaware of which allocation, LAIV H7N9 or matched placebo, is received; study vaccine and placebo will be masked. Subjects will be carefully monitored for adverse reactions while in the isolation unit.

All subjects will remain in the isolation unit for at least 6 days after receipt of study vaccine or placebo. Nasal swabs will be collected daily while subjects are in isolation to test for presence of influenza virus shed in the nasal passage. Any subject exhibiting conjunctivitis will also have a conjunctival swab collected on the day of appearance of the sign. Any subject exhibiting influenza A virus shedding, as determined by real-time RT-PCR positivity on a nasal swabs specimen, in the 2 days prior to each planned discharge day after each dose (Days 5 or 6 or Days 33 or 34) will be kept in the isolation until PCR-diagnosis results confirm that no influenza virus is present in a tested clinical specimens for at least two consecutive days.

Any subject still exhibiting evidence of influenza virus shedding in a nasal swabs on Days 5 or 6 or Days 33 or 34 post-administration with each dose will be placed on approved influenza antiviral (oseltamivir) treatment at the standard dose for treatment of 75 milligrams (mg) twice a day for a course of 5 days.

After discharge from the isolation unit, subjects will complete diary cards for AEs and use of concomitant medications. Subjects will return to the isolation unit at four weeks (Day 28) after administration of dose one of study vaccine or placebo. At that time, similar procedures will be used for admittance to the isolation unit, for receipt of dose two of study vaccine or placebo and for isolation and follow-up, with the additional procedure of review of interim histories (and diary cards) since first discharge after dose one.

After second discharge from the isolation unit, subjects will again complete diary cards for AEs and use of concomitant medications. Subjects will then return to the study center at four weeks (Day 56) after administration of dose two of study vaccine or placebo for their study visit. Interim histories (and diary cards) will again be reviewed and blood and nasal wick specimens will be collected. Women will also undergo a final pregnancy screen.

For assessment of safety, subjects will be observed for two hours after each administration of study vaccine or placebo. Twice daily (early morning and late afternoon) examination will be also used to assess reactions for 6 days after each administration of study vaccine or placebo. ENT examination and examination by neurologist will also occur once per day on Days 6, 28, 34 and 56. Subjects will complete diary cards for unsolicited AEs from the day of each discharge until return to the isolation unit for dose two (at Day 28) or until return to the study center for the final study visit at four weeks post dose two (at Day 56). To assess safety, blood and urine specimens will also be collected on days 3, 6, 28 (prior to administration of dose two of study vaccine or placebo), days 31, 34 and 56 for testing by routine biochemical and hematological blood tests and urinanalysis respectively. On the 0th, 3rd and 31st days of the study, instrumental examinations will be carried out (ECG, echocardiogram, and spirometry with the assessment of respiratory function). In order to assess late adverse events, volunteers will remain under observation for 6 months after the second vaccination (28th day of the study) with monthly monitoring of their health condition by telephone.

For the evaluation of mucosal IgA antibody, nasal wick and saliva specimens will be collected on Day 0 (prior to administration of dose one of study vaccine or placebo), on Day 28 (prior to administration of dose two of study vaccine or placebo) and on Day 56. For the evaluation of serum antibodies (by HAI, microneutralization and IgA and IgG ELISA), serum specimens will be collected on Day 0 (prior to administration of dose one of study vaccine or placebo), on Day 28 (prior to administration of dose two of study vaccine or placebo) and on Day 56. To study virus infectivity (by isolation in embryonated chicken eggs) and viral genetic stability (by molecular sequencing of any isolated virus), nasal swab specimens will be taken on Days 1, 2, 3, 5, 6, 29, 30 and 31. To assess priming and stimulation of cytotoxic T lymphocytes and other cytokine indicators, whole blood for isolation of PBMCs will be collected on Days 0 (prior to administration of dose one of study vaccine or placebo), on Day 6 (prior to discharge from isolation unit), on Day 28 (prior to administration of dose two of study vaccine or placebo), and on Day 56.

The primary study hypothesis is that two doses of cold-adapted, live monovalent (H7N9) influenza vaccine will be safe in healthy adults.

Observed proportions of subjects exhibiting reactions, adverse events and clinical chemistry anomalies, as well as proportions of subjects seroconverting or seropositive for influenza antibodies using various methods, will be estimated with 95% confidence intervals. Geometric mean titers (GMTs) will be estimated with 95% confidence intervals. The study will be primarily evaluated based on the exact two-sided 95% confidence interval of the percentage of vaccine recipients experiencing vaccine-related serious adverse events within 28 days of any dose.

ELIGIBILITY:
Inclusion Criteria:

* Legal male or female adult 18 through 49 years of age at the enrollment visit.
* Literate and willing to provide written informed consent.
* A signed informed consent.
* Free of obvious health problems, as established by the medical history and screening evaluations, including physical examination.
* Capable and willing to complete diary cards and willing to return for all follow-up visits
* Willing to comply with the rules of the isolation unit (including willing and able to take oseltamivir influenza antiviral medication, should that be recommended by a study physician).
* For females, willing to take reliable birth control measures through day 56.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until four weeks after study completion.
* Practice of nasal irrigation on a regular basis within the past six months or has engaged in nasal irrigation within two weeks prior to enrollment.
* Recent history of frequent nose bleeds (more than 5 within the past year).
* Clinically relevant abnormal paranasal anatomy.
* Recent history (within the past month) of rhino or sinus surgery, or surgery for any traumatic injury of the nose.
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Other acute illness at the time of study enrollment.
* Receipt of immune globulin or other blood products within three months prior to study enrollment or planned receipt of such products during the period of subject participation in the study.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, 0.5 mg per kg per day; topical steroids are allowed, exclusive of nasal.)
* Participation in any previous trial of any H7 or H5 containing influenza vaccine.
* History of bronchial asthma.
* Hypersensitivity and allergy reactions after previous administration of any vaccine.
* History of wheezing after past receipt of any live influenza vaccine.
* Other AE following immunization (body temperature more than 40°C, collapse, non-febrile seizures, anaphylaxis), at least possibly related to previous receipt of any vaccine (not only influenza).
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein.
* Seasonal (autumnal) hypersensitivity to the natural environment.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, metabolic, neurologic, psychiatric or renal functional abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives. Subjects with physical examination findings or clinical laboratory screening results which would be graded 2 or higher on the AE severity grading scale (see Attachments) will be excluded from entry into the study and will be excluded from receipt of dose two of study vaccine or placebo.
* History of leukemia or any other blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressive or immunodeficient condition of any kind, including HIV infection.
* Known chronic HBV or HCV infection.
* Known tuberculosis infection or evidence of previous tuberculosis exposure according to anamnesis and/or available medical records.
* History of chronic alcohol abuse and/or illegal drug use.
* Claustrophobia or sociophobia according to anamnesis and/or available medical records.
* Pregnancy or lactation. (A negative pregnancy test will be required before administration of study vaccine or placebo for all women of childbearing potential.)
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if he/she participates in the study or would interfere with the evaluation of the study objectives.
* Allergic, including anaphylactic, reactions to the introduction of any vaccines in the subject's medical history (not only flu vaccine).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-03 (Estimated); Primary Completion 2019-06-03 (Estimated); Study Completion 2019-07-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Immediate reactions | 2 hours
  Proportion of subjects experiencing immediate reactions (related or not related to the study) occuring within two hours of administration of any dose, measured as observed by study staff or reported by the subject to study staff
Number of Participants with Solicited adverse events | greater than two hours after administration of any dose of study vaccine or placebo through 6 days following any dose
  Proportion of subjects experiencing adverse events (related or not related to the study) commonly associated with intranasal vaccination (solicited local and systemic reactions) occurring greater than two hours after administration of any dose of study vaccine or placebo through 6 days following any dose, measured as observed by study staff or reported by the subject to study staff.
Number of Participants with Changes from baseline in laboratory findings and instrumental tests (ECG, echocardiogram, and spirometry) | Days 3, 6, 31 and 34
  Proportion of subjects experiencing all other adverse events (including unsolicited events) occurring during the 6 days following any dose, measured as observed by study staff or reported by the subject to study staff. This includes abnormal laboratory findings from blood specimens and urinalysis collected on Days 3, 6, 31 and 34; IgE level data for Days 0, 3, 28, and 56, as well as instrumental test data (ECG, echocardiogram, and spirometry) on the third day after each vaccination.
Number of Participants with Serious adverse events (SAEs) | 4 weeks of receipt of any dose
  Proportion of subjects experiencing all serious adverse events (SAEs) occurring within 4 weeks of receipt of any dose, as observed by study staff, reported by the subject to study staff, or noted by the subject on a diary card. This includes abnormal laboratory findings from blood specimens collected on Days 28 (pre-vaccination) and 56.

SECONDARY OUTCOMES:
Number of Participants with Immune responses | Days 0, 3, 28, and 56
  Immune responses was parameterized as the proportion of subjects with at least a four-fold rise after each dose from baseline or as the mean titer after each dose in any of the following:
  * Serum hemagglutination-inhibition antibodies
  * Serum neutralizing antibodies using microneutralization assay
  * Serum immunoglobulin class A (IgA) and class G (IgG) antibodies using enzyme-linked immunosorbent assay (ELISA)
  * Secretory IgA antibodies from the nasal mucosa detected in nasal wick specimens using ELISA
  * Secretory IgA antibodies detected in saliva specimens using ELISA
Number of Participants with Virus shedding at Days 0-6 after each dose | Days 0-6 after each dose
  Virus shedding will be parameterized as the proportion of subjects shedding virus [detected by real-time reverse transcriptase polymerase chain reaction (rRTPCR) in nasal or conjunctival swabs] at any time-point. Shedding data will be reported for every subject at every measured time-point.
Number and name of mutations leading to any loss of attenuation phenotype of the vaccine virus (genetic stability) | Days 0-6 after each dose
  The influenza virus will be isolated in chicken embryos from all PCR influenza A positive nasal or conjunctival swabs collected during 6 days after any vaccine dose. Molecular characterization of any shed virus will be reported with sequence details of any loss of attenuation mutations.

OTHER OUTCOMES:
Cellular immune responses (cytokines and T-cells) | Days 0, 28, and 56
  Cellular immune responses (cytokines and T-cells) will be measured using isolated peripheral blood mononuclear cells tested by flow cytometry and ELISPOT techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Larisa G Rudenko, MD, PhD, DSc, Study Chair — Institute of Experimental Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiseleva I, Isakova-Sivak I, Stukova M, Erofeeva M, Donina S, Larionova N, Krutikova E, Bazhenova E, Stepanova E, Vasilyev K, Matyushenko V, Krylova M, Galatonova J, Ershov A, Lioznov D, Sparrow EG, Torelli G, Rudenko L. A Phase 1 Randomized Placebo-Controlled Study to Assess the Safety, Immunogenicity and Genetic Stability of a New Potential Pandemic H7N9 Live Attenuated Influenza Vaccine in Healthy Adults. Vaccines (Basel). 2020 Jun 10;8(2):296. doi: 10.3390/vaccines8020296. PMID 32532097